CLINICAL TRIAL: NCT01841411
Title: Studying the Role of N-Acetyl Cysteine Either Alone or in Combination With Metronidazole in Treatment of Bacterial Vaginosis
Brief Title: Role of N-Acetylcysteine in Treatment of Bacterial Vaginosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Heba Ahmed Mohamed, principal investigator, Minia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Microbiology2013
Record Dates: First submitted 2013-03-15; First posted 2013-04-26 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Bacterial Vaginosis
Keywords: bacterial vaginosis, recurrence, N-Acetyl cysteine
MeSH Terms: conditions — Vaginosis, Bacterial; Recurrence | interventions — Acetylcysteine; Metronidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Metronidazole + N-Acetyl cysteine (Experimental): the second patient group will use NAC sachets containing 200 mg as a vaginal douche once daily plus oral metronidazole 500 mg twice daily for 7 days
  Interventions: Drug: Metronidazole + N-Acetyl cysteine
- N- Acetyl cysteine (Experimental): the third patient group will use NAC sachets containing 200 mg as a vaginal douche only without taking metronidazole
  Interventions: Drug: N-Acetyl cysteine
- Metronidazole (Active Comparator): the first group of patients will take oral metronidazole 500 mg twice daily for a week
  Interventions: Drug: metronidazole

INTERVENTIONS:
Drug: N-Acetyl cysteine — N-Acetyl cysteine is a pharmaceutical drug and nutritional supplement,it is a derivative of the natural amino acid cysteine, from which it differs by virtue of the introduction of an acetyl group on the nitrogen atom of the amino terminal.It is used mainly as a mucolytic and in management of paracetamol overdose. It has been observed that N-acetyl cysteine has shown good properties in terms of combating bacterial infections. In particular, it has been observed that NAC presents good activity in terms of inhibiting bacterial adhesion and in dissolving the biofilm matrix.
  Other Names: Acetyl cistein
  Arms: N- Acetyl cysteine
Drug: Metronidazole + N-Acetyl cysteine — Metronidazole is an antibiotic effective against anaerobic bacteria and certain parasites.It can be used in treatment of vaginal infections such as trichomoniasis and bacterial vaginosis N-Acetyl cysteine is a pharmaceutical drug and nutritional supplement, It is used mainly as a mucolytic and in management of paracetamol overdose. It has been observed that N-acetyl cysteine has antibacterial and antibiofilm activities
  Other Names: Flagyl, Acetyl cistein
  Arms: Metronidazole + N-Acetyl cysteine
Drug: metronidazole — Metronidazole is an antibiotic effective against anaerobic bacteria and certain parasites.It can be used in treatment of vaginal infections such as trichomoniasis and bacterial vaginosis in treatment of bacterial vaginosis, it can be used in treatment of bacterial vaginosis either in a dose of 500 mg twice daily or 250 mg three times daily for seven days
  Other Names: Flagyl
  Arms: Metronidazole

SUMMARY:
N-Acetyl cysteine (NAC) is an amino acid with strong antioxidant, mucolytic and antibacterial properties, and is produced within the human body.Its effect in biofilms has been tested in several bacteria. Biofilms have recently been observed in 90% of subjects with bacterial vaginosis (BV) with Gardnerella vaginalis being the predominant species. Although a wide range of antimicrobial agents are currently available, treatment options for controlling BV are still limited. Furthermore, the number of relapses are increasing and require alternative treatments. This study is aiming to evaluate the role of NAC in treatment of BV and prevention of recurrence.

DETAILED DESCRIPTION:
Bacterial vaginosis (BV) is the most frequent diagnosis made in women with lower genital tract symptoms. It has recently been observed that 90% of subjects with BV show the growth of bacteria in the form of biofilms,and that Gardnerella vaginalis was the predominant species. The propensity of G. vaginalis to form biofilm is clinically relevant because this form of growth allows it to tolerate higher concentrations of certain antibiotics, thus increasing the possibility of recurrent BV even after apparently curative therapy. So new treatment strategies must be used to insure complete cure and prevent recurrence. NAC is an amino acid with strong antioxidant, mucolytic and antibacterial properties, and is produced within the human body.Its effect in biofilms has been tested in several bacteria.

This study aims to test the efficacy of NAC in treatment of BV either alone or in combination with the traditionally used metronidazole. Also the effect of using NAC in prevention of recurrence of BV will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* patients complaining bacterial vaginosis and proved to have BV using standard diagnostic methods for BV
* patients with age between 20-50

Exclusion Criteria:

* Virgins and menstruating patients.
* Recent douching or sexual intercourse.
* Use of systematic or vaginal antimicrobial therapy or any vaginal suppositories or drugs.

All patients will sign a written consent before starting the treatment

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
recovery of BV | one week
  Vaginal swabs from all patients will taken and smears will be gram stained, examined and evaluated according to Nugent scoring system afetr one week of treatment. The patient will be considered recovered if she have Nugent score of 0-3.

SECONDARY OUTCOMES:
prevention of recurrence | 3 months
  patients who recovered after treatment will be asked for symptoms of recurrence of bacterial vaginosis and vaginal smears will be evaluated according Nugent scoring system after one month, two months and three months from the date of the end of initial treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed R El-Adawy, Professor, Study Chair — Minia university hopital of gynecology and obstetrics; Heba A Mohamed, MSc, Principal Investigator — Minia University
Locations (1):
- Minia university hospital for gynecology and obstetrics, Minya, Egypt